CLINICAL TRIAL: NCT04328103
Title: Combining Electrophysiological, Behavioral and Psychological Measures to Target Mechanisms of Emotion Processing and Regulation During Cognitive Behavior Therapy in Depression
Brief Title: Mechanisms of Emotion Regulation Underlying Successful CBT in Depression
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jürgen Kayser, PhD, Research Scientist / Professor of Clinical Neurobiology, New York State Psychiatric Institute
Other Study IDs: 6559R
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder
Keywords: Cognitive Behavioral Therapy (CBT); Motivated Attention; Psychological Mindedness; Mindfulness; Visual Half-Field paradigm; Dichotic Listenting; Emotion Recognition Task; Left Ear Advantage (LEA); Emotion Regulation; Event-Related Potential (ERP); Meta-Cognitive Processes
MeSH Terms: conditions — Depressive Disorder, Major; Emotional Regulation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitive Behavior Therapy (CBT): Following established procedures at the Depression Evaluation Service (DES) at New York State Psychiatri Institute (NYSPI), 12 sessions of individual manual-driven CBT (Emery, 2000) will be conducted by highly trained master degree clinicians.
  Interventions: Behavioral: Cognitive Behavior Therapy (CBT)
- Nonspecific Supportive Therapy (PBO): As a non-CBT intervention that includes warmth, genuineness and empathy (Linde et al., 2011), nonspecific supportive therapy (PBO) will be administered in a parallel format to CBT, also consisting of 12 individual sessions.
  Interventions: Behavioral: Nonspecific Supportive Therapy (PBO)

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy (CBT) — Following established procedures at the DES at NYSPI, 12 sessions of individual manual-driven CBT (Emery, 2000) will be conducted by highly trained master degree clinicians.
  Groups: Cognitive Behavior Therapy (CBT)
Behavioral: Nonspecific Supportive Therapy (PBO) — As a non-CBT intervention that includes warmth, genuineness and empathy (Linde et al., 2011), nonspecific supportive therapy (PBO) will be administered in a parallel format to CBT, also consisting of 12 individual sessions.
  Groups: Nonspecific Supportive Therapy (PBO)

SUMMARY:
This research aims to elucidate mechanisms through which change occurs during cognitive behavior therapy (CBT) for depression. Assessing meta-cognitive processes of self-knowledge (top-down), electrophysiological and behavioral correlates of emotion processing (bottom-up), and their relation to treatment outcome will provide new insights into the mechanisms of emotion regulation deficits in depression. It will also contribute toward the clinical goal of identifying patients who may benefit most from CBT for unipolar depression.

DETAILED DESCRIPTION:
This R21 application aims to clarify the neurobiological mechanisms by which change occurs during cognitive behavior therapy (CBT) for major depressive disorder (MDD). This hypothesis-driven study will explore the association between the psychological constructs of psychological mindedness (PM) and mindfulness (M) during the time course of CBT for MDD, and its relationship to electrophysiological and behavioral measures of automatic (i.e. stimulus-driven or bottom-up) emotion processing. This objective is motivated by the following rationale: PM and M represent different meta-cognitive processes of self-knowledge deemed critical for emotion regulation (ER) and CBT success. Event-related potentials (ERPs) to salient affective pictures reflect different stages of motivated attention. Using advanced analytic EEG techniques, we have linked these stages to the hierarchical activation of 'emotional' brain regions along the occipitotemporal ventral stream, ranging from preconscious stimulus categorization (right secondary visual cortex, right temporoparietal junction) to conscious appraisal (posterior cingulate cortex, ventromedial cortex). Importantly, blunted ERP responses to emotionally-arousing stimuli have been observed in clinical depression, and hypoactivation of right temporoparietal and dorsolateral prefrontal regions normalize after successful antidepressant or electroconvulsive treatment. A dichotic emotion recognition test, which provides an auditory measure of bottom-up emotion processing in form of a left ear (right hemisphere) advantage for recognizing the emotional intonation of speech patterns, has revealed behavioral deficits in MDD patients. Moreover, an increased right ear advantage for verbal stimuli (left hemisphere) is seen in CBT responders. Employing a sample of 60 MDD patients randomly assigned to CBT or nonspecific supportive therapy (placebo), we will obtain psychological, electrophysiological, behavioral and clinical outcome measures of response to 12 weeks of CBT in a pre-post treatment design to determine: (1) when and where in the brain automatic emotion processing is altered by CBT; (2) if changes in emotional responding are moderated or mediated by meta-cognitive processes of self-knowledge; and, (3) if these measures, alone or in combination, have promise as markers of CBT treatment response. Existing ERP and behavioral data for healthy adults (HC) obtained using the same experimental protocols will provide normative (yardstick) data. This study brings together experienced clinical psychologists and psychiatrists doing treatment and research in depression with investigators having expertise in affective neuroscience and electrophysiological studies in MDD. It will provide a critical new step for outlining the affective-cognitive and neurophysiological mechanisms of ER by which change through CBT occurs. Apart from their theoretical relevance, the findings of this project will also aid in developing novel and more targeted interventions and in identifying patients who may benefit most from CBT for unipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65
* right-handed
* be able to speak English well enough to comprehend and comply with protocol requirements
* recruited to achieve equal gender representation (i.e. about half male) in both treatment arms
* medically healthy individuals will be included as MDD patients if they:

  1. meet DSM-5 criteria for a current MDD episode based on a structured clinical interview (SCID);
  2. score greater or equal to 13 on the Beck Depression Inventory (BDI-II)
  3. score greater or equal to 14 on the Hamilton Rating Scale for Depression (HRSD)

Exclusion Criteria:

* Participants are excluded for any of the following reasons or DSM-5 criteria:

  1. substance abuse or dependence (including alcohol) in last 6 months;
  2. positive toxicology screen as determined by blood/urine testing (e.g. thyroid dysfunction, street drug use);
  3. history of schizophrenia or other current psychotic disorder;
  4. MDD with psychotic or catatonic features;
  5. Bipolar I, II Affective Disorder;
  6. Organic Mental Disease;
  7. significant suicidal ideation with a plan and intent, also assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS), that cannot be managed safely as an outpatient, or homicidal ideation (suicidality monitored throughout study);
  8. a primary diagnosis of panic disorder, obsessive-compulsive disorder, psychogenic pain disorder, anorexia/bulimia, or any unstable medical condition;
  9. any recent (less than or equal to 12 mos) history of CBT (as determined during an in-person interview);
  10. prior seizure disorder, significant head trauma or other neurological disorders;
  11. lack of capacity to give informed consent;
  12. received psychotropic medication, over-the-counter antidepressant, or any non-CBT intervention (e.g. deep breathing, meditation/mindfulness, psychotherapy - except for minimal supportive nonspecific therapy PBO) for at least 1 month prior to recruitment (3 months for fluexetine);
  13. hearing loss (>30 dB in either ear) or hearing asymmetry (>10 dB across ears) assessed via standard audiogram

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Right-handed MDD patients (N = 60; Beck Depression Inventory [BDI] > 12, Hamilton Rating Scale for Depression [HRSD] > 13), aged 18 to 65 (~half male), recruited through the Depression Evaluation Service at NY State Psychiatric Institute (NYSPI)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
HRSD slope | 12 weeks or up to 12 weeks
  17-item Hamilton Rating Scale for Depression (HRSD); standard clinical instrument (Hamilton, 1960) to assess symptom severity in major depressive disorder (MDD); interpretation: < 7 = absence or remission of depression; 7-17 = mild depression; 18-24 = moderate depression; > 25 = severe depression;
  HRSD rate of symptom change over time (slope); to obtain a continuous measure of treatment outcome, we will employ a mixed-effects model for all HRSD ratings to compute estimates of each patient's rate of symptom change over time (slope of HRSD scores; Petkova et al 2017)
BDI slope | 12 weeks or up to 12 weeks
  Beck Depression Inventory (BDI-II); standard clinical instrument (Beck 1966) to assess symptom severity in depression; interpretation: < 14 = minimal range; 14-19 = mild depression; 20-28 = moderate depression; 29-63 = severe depression;
  BDI-II rate of symptom change over time (slope); To obtain a continuous measure of treatment outcome, we will employ a mixed-effects model for all BDI ratings to compute estimates of each patient's rate of symptom change over time (slope of BDI scores; Petkova et al 2017)
N2 sink (pre) | pre-treatment, at baseline
  N2 sink (ERP, Emotional Hemifield Task); early (212 ms peak latency) emotional ERP LPP subcomponent derived from combined CSD-tPCA approach (Kayser et al 2016, 2017) reflecting asymmetrical neuronal sources involving striate and prestriate cortex in the occipital lobe, with a maximum activation in the right middle temporal gyrus
N2 sink (post) | post-treatment, after about 12 weeks
  N2 sink (ERP, Emotional Hemifield Task); early (212 ms peak latency) emotional ERP LPP subcomponent derived from combined CSD-tPCA approach (Kayser et al 2016, 2017) reflecting asymmetrical neuronal sources involving striate and prestriate cortex in the occipital lobe, with a maximum activation in the right middle temporal gyrus
P3 source (pre) | pre-treatment, at baseline
  P3 source (ERP, Emotional Hemifield Task); mid-latency (385 ms peak latency) emotional ERP LPP subcomponent derived from combined CSD-tPCA approach (Kayser et al 2016, 2017) reflecting neuronal sources involving medial parietal lobe, with a maximum activation in the posterior cingulate cortex
P3 source (post) | post-treatment, after about 12 weeks
  P3 source (ERP, Emotional Hemifield Task); mid-latency (385 ms peak latency) emotional ERP LPP subcomponent derived from combined CSD-tPCA approach (Kayser et al 2016, 2017) reflecting neuronal sources involving medial parietal lobe, with a maximum activation in the posterior cingulate cortex
CP source (pre) | pre-treatment, at baseline
  CP source (ERP, Emotional Hemifield Task); late (630 ms peak latency) emotional ERP LPP subcomponent derived from combined CSD-tPCA approach (Kayser et al 2016, 2017) reflecting bilateral generator sources within the temporal lobe, with a maximum activations in uncus and the inferior temporal area
CP source (post) | post-treatment, after about 12 weeks
  CP source (ERP, Emotional Hemifield Task); late (630 ms peak latency) emotional ERP LPP subcomponent derived from combined CSD-tPCA approach (Kayser et al 2016, 2017) reflecting bilateral generator sources within the temporal lobe, with a maximum activations in uncus and the inferior temporal area
LEA ERT (pre) | pre-treatment, at baseline
  LEA ERT (dichotic listing behavior, Emotional Recognition Task); measures extent of right hemisphere dominance or left ear advantage (LEA) for recognizing prosody during a dichotic emotional recognition task (Bruder et al 2016)
LEA ERT (post) | post-treatment, after about 12 weeks
  LEA ERT (dichotic listing behavior, Emotional Recognition Task); measures extent of right hemisphere dominance or left ear advantage (LEA) for recognizing prosody during a dichotic emotional recognition task (Bruder et al 2016)

SECONDARY OUTCOMES:
REA Fused Words (pre) | pre-treatment, at baseline
  REA Fused Words (dichotic listing behavior); measures extent of left hemisphere dominance or right ear advantage (REA) for verbal processing (Bruder et al 1997, 2017)
REA Fused Words (post) | post-treatment, after about 12 weeks
  REA Fused Words (dichotic listing behavior); measures extent of left hemisphere dominance or right ear advantage (REA) for verbal processing (Bruder et al 1997, 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Kayser, PhD, Principal Investigator — NYSPI/RFM/CU; Ronit Kishon, PhD, Principal Investigator — NYSPI/RFM/CU
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The institution and PIs will adhere to the NIH Data Sharing Policy (Notice of Data Sharing Policy for the National Institute of Mental Health NOT-MH-19-033). Accordingly, we will deposit de-identified individual raw and analyzed data (primary and secondary outcome measures) from experiments involving human subjects into the NIMH Data Archive (NDA) infrastructure (i.e., for all data for which we will obtain informed consent). Raw data will be submitted to NDA every 6 months and include demographic, self-report, clinical, and EEG, following NDA Harmonization Standards (i.e., for clinical/phenotypic data and neuro-signal recordings) and using NDA GUIDs. These submissions will undergo validations and other quality control checks as the data are deposited.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available 12 months after end of NIMH funding (06/30/2023).
Access Criteria: Data will be available through the NIMH Data Archive (NDA depositiory).
URL: https://nda.nih.gov/